CLINICAL TRIAL: NCT03279562
Title: Patient Driven Recovery With Nalmefene and Coaching
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: First Pavlov State Medical University in St. Petersburg, Russia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1610018492
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Opioid-use Disorder; Harmful; Use, Alcohol
MeSH Terms: conditions — Opioid-Related Disorders | interventions — nalmefene

STUDY DESIGN:
Intervention Model Description: Pilot, open label, non-randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nalmefene and recovery coaching (Experimental): Nalmefene prescribed for daily ingestion during the first 3 months of treatment; patients who maintain a successful recovery during the first 3 months of treatment will be offered an option to take Nalmefene on as needed basis, always before encountering situations or circumstances with heightened risk of alcohol or opioid use
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Nalmefene — Educational and behaviorally oriented drug counseling
  Other Names: Recovery coaching

SUMMARY:
In collaboration with the First Pavlov State Medical University in St. Petersburg, Russia, we are proposing a pilot, open label, non-randomized clinical trial to evaluate the safety, feasibility, acceptability, and preliminary efficacy of treatment for alcohol and opioid use disorders combining Nalmefene and recovery coaching (educational and behaviorally oriented drug counseling). The proposed pilot study will also be used to further develop and refine the recovery coaching/counseling intervention and to train additional cadre of clinicians and researchers in St. Petersburg, Russia.

DETAILED DESCRIPTION:
The specific aims and hypotheses of the proposed study are as follows:

Specific Aim 1: To evaluate the safety, feasibility, acceptability, and preliminary efficacy of treatment of alcohol and opioid use disorders combining Nalmefene and recovery coaching for rehabilitation of detoxified opioid dependent individuals in Russia.

Specific Aim 2: To further develop and refine the recovery coaching/counseling intervention and to train additional cadre of clinicians and researchers in St. Petersburg, Russia.

ELIGIBILITY:
Inclusion Criteria:

* individuals who meet DSM IV criteria for opioid dependence, who use street methadone (the main, most frequently used street opioid in Saint Petersburg, Russia) by intravenous injections, who have a history of alcohol use disorder or high risk alcohol use, who successfully completed inpatient, medically supervised detoxification, who are seeking a rehabilitation treatment following detoxification, and who pass a naloxone challenge (indicating the current lack of physiological dependence on opioids)

Exclusion Criteria:

* current suicide or homicide risk; current psychotic disorder or major depression; inability to understand the consent form or assessments; pregnancy; acute medical conditions requiring medical treatment, co-occurring dependence/abuse of other drugs including alcohol, benzodiazepines, or amphetamine type stimulants (ATS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Duration of abstinence from illicit opioids | Past 30 days
  Days of abstinence from illicit opioids, based on urine tests and self-report

SECONDARY OUTCOMES:
Treatment retention | 6 months
  Duration of treatment participation, number of days in treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, Department, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No